CLINICAL TRIAL: NCT02482545
Title: Breakfast Meal Replacement Use on Body Composition and Health-related Quality of Life in Overweight Men and Women: a Randomized Controlled Trial
Brief Title: Breakfast Meal Replacement
Acronym: MRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Abbie Smith-Ryan, PhD, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 15-0543
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Body Composition, Beneficial; Basal Metabolic Rate; Satiety; Overweight; Obese
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breakfast Meal Replacement (Experimental): Once daily of a powdered meal replacement (high fat, high protein) will be consumed, mixed with water, at breakfast.
  Interventions: Dietary Supplement: Meal replacement
- Control (No Intervention): No placebo or intervention

INTERVENTIONS:
Dietary Supplement: Meal replacement
  Arms: Breakfast Meal Replacement

SUMMARY:
Purpose: To evaluate the effects of replacing breakfast with a high protein, high fat, high fiber meal replacement in overweight individuals, on body composition.

Participants: Healthy, overweight and obese individuals (ages 18-45 yrs) with no history of disease. Procedures (methods): In a randomized control intervention, subjects will complete 5 different testing sessions (pre-screening, 2 baseline testing sessions, and 2 post testing sessions) as well as an 8 week intervention period. Pre-screening will include written informed consent, health history questionnaire, nutrition analysis, and baseline anthropometric measures. Baseline testing will be split into two sessions and include measurements of resting metabolic rate (RMR), body composition, blood and saliva hormones, mood, satiety, and health related quality of life questionnaires, and a cardiorespiratory fitness assessment.

Subjects will be randomly assigned to treatment (8 week supplementation with meal replacement to be taken at breakfast) and control groups (continue normal eating habits) with 4 electronic correspondences throughout the supplementation period. All measures will be repeated in two post-testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Overweight Men and Pre-Menopausal Women
* Participant agrees to maintain usual activity lifestyle
* Participant has a body mass index of ≥ 28 (men) and ≥25 (women) kg/m2 and/or %body fat of ≥ 25%
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire (diabetes, heart disease, kidney disease, cancer, thyroid disorder, etc).
* Participant agrees to abstain from smoking, caffeine, tobacco, and alcohol before testing days
* Participant has stated a goal of losing weight or improving body composition

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders (i.e. anything influencing exercise ability).
* Participant is using, or has used one of the following dietary supplements within 8 weeks prior to enrollment: Meal replacement shakes, Whey Protein, Beta-alanine, Creatine, beta-hydroxy beta methylbutyrate, Carnosine or Taurine
* Participant has lost or gained greater than ten pounds within the previous 3 months
* Participant is in, or has participated in another clinical trial within 4 weeks prior to enrollment
* Participant had or currently has a self-identified eating disorder
* Participant is pregnant or plans to become pregnant during the duration of the study
* Participant has a known allergy or sensitivity to any ingredient in the test product or placebo (determined from health history questionnaire)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Fat Mass measured from multi-compartment (4C) model | 0 to 8 weeks

SECONDARY OUTCOMES:
Change in lean mass measured from multi-compartment (4C) model | 0 to 8 weeks
Change in percent body fat measured from multi-compartment (4C) model | 0 to 8 weeks
Change in resting metabolic rate using indirect calorimetry | 0 to 8 weeks
Change in respiratory exchange ratio using indirect calorimetry | 0 to 8 weeks
Change in total leptin concentrations from blood sample analysis | 0 to 8 weeks
Change in LDL from blood sample analysis | 0 to 8 weeks
Change in triglycerides from blood sample analysis | 0 to 8 weeks
Change in insulin from blood sample analysis | 0 to 8 weeks
Change in visceral fat from ultrasonography | 0 to 8 weeks
Change in satiety via questionnaire | 0 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, Principal Investigator — University of North Carolina
Locations (1):
- Applied Physiology Laboratory, Chapel Hill, North Carolina, United States